CLINICAL TRIAL: NCT05990556
Title: Research on the Safety and Efficacy of Blocking Dural Blood Supply in Glioblastoma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhang Nu, Discipline Leader of Neurosurgery department, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZNu
Record Dates: First submitted 2023-08-07; First posted 2023-08-14 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Glioblastoma; Meningeal Arteries
Keywords: glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: Interventional single-arm studies, no grouping.
  1 Randomize groupings 1.1 Method for generating random sequence assignments This study is a real-world study, it is planned to include 20 patients as a case, there is no need for random sequence and blinded allocation before intervention, the patient's condition, experimental purpose, experimental method and possible risks are informed before surgery, and the patient chooses whether to undergo preoperative interventional surgery to block bilateral meningeal blood supply.
  1.2 Randomly assigned hiding This is a real-world study that intends to include three patients as individual cases without random sequencing prior to intervention and therefore does not involve allocation concealment.
Masking Description: Blinding and unblinding This is a real-world study that intends to include three patients as case studies without blinding prior to intervention and therefore does not involve blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional procedure to block bilateral meningeal blood supply (Experimental)
  Interventions: Procedure: interventional procedure to block bilateral meningeal blood supply

INTERVENTIONS:
Procedure: interventional procedure to block bilateral meningeal blood supply — The embolic agent used in bilateral meningeal blood supply occlusion through interventional surgery is Onyx glue ("liquid embolic system"). After the location of bilateral middle meningeal artery was determined by femoral artery puncture angiography, SL-10 was sent to the opening of bilateral middle meningeal artery through guiding catheter, and Onxy glue was used to block the bilateral middle meningeal artery. The standard of embolization was that the middle meningeal artery was not seen and Onyx glue was not diffused to the petrous branch of the middle meningeal artery. In order to avoid dangerous anastomotic branches and complications, attention should be paid to superselecting the middle meningeal artery and slowly injecting Onyx glue during the operation. After embolization of the middle meningeal artery by interventional surgery, glioblastoma was removed immediately under the guidance of multimodal imaging.

SUMMARY:
Glioblastoma is the most common primary malignancy of the central nervous system with a very poor prognosis. Most of the immunotherapies that have made significant breakthroughs in the treatment of other tumors in recent years are unsatisfactory in the application of glioblastoma, which is mainly inseparable from the highly inhibitory immune microenvironment formed by the latter. Therefore, how to change this "immune desert" and better activate immune effector cells to play an anti-tumor effect is currently a hot spot in glioma immune research. In recent years, there has been continuous research support that the myeloid cells of the central nervous system are partly derived from the bone marrow of the skull, and there is a special channel connection between the skull and the dura mater, through which immune cells can be transported. This suggests that some of the tumor-associated macrophages recruited in the glioblastoma microenvironment may be passed through the dura mater. In previous animal experiments, we blocked the main blood supply to the dura mater by ligating the bilateral external carotid arteries of mice, cutting off the potential supply of dura mater to suppressor myeloid cells in the lesion. The results showed that after ligation of bilateral external carotid arteries, the survival period of tumor-forming mice was significantly prolonged and the prognosis was improved. The proportion of myeloid cells in the tumor microenvironment of mice decreased significantly, and the expression of tumor suppressor molecules such as arginase Arg1 decreased, indicating that the improvement of mouse prognosis was closely related to the proportion and phenotypic changes of myeloid cells after dural blood supply blockade. The meningeal lymphatic system of the human central nervous system has been shown to be an important part of the immune system, while the external carotid artery system, the main source of blood supply to the dura, carries abundant immune cells that ooze out to the dura mater through the endothelial window hole of the dural blood vessel, which is an important source of dural immune cells. In the glioblastoma immune microenvironment, the source of immune cells includes dural branches from the external carotid artery system in addition to branches of the internal carotid artery system. Therefore, for patients diagnosed with glioblastoma, this study involves embolization of the dural branch of the external carotid artery system (bilateral middle meningeal artery) to block the dural blood supply before craniotomy. At the same time, microsurgery under multimodal image navigation was used to remove the tumor. It is expected to be effective in reducing the proportion of myeloid suppressor cells in the tumor microenvironment, slowing the growth rate of residual tumor cells, and prolonging the tumor-free progression and survival of patients.

ELIGIBILITY:
Inclusion Criteria:

* Imaging or needle biopsy pathologically diagnosed as glioblastoma
* Patients have not previously received radiotherapy, chemotherapy and other treatment modalities for intracranial lesions
* There are no related contraindications such as neurovascular intervention and craniotomy

Exclusion Criteria:

* The patient's initial imaging diagnosis was glioblastoma, and the postoperative pathology confirmed nonglioblastoma
* The patient has other underlying medical conditions that affect survival time
* The patient had other underlying medical conditions that affected follow-up or quality of life assessment
* Patients do not have the above exclusion criteria and refuse to participate in clinical trials after informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-11 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival period | 15 months
  The overall survival of enrolled patients was compared with the overall survival reported in the literature

SECONDARY OUTCOMES:
Postoperative recurring time | 3-6 months
  The Postoperative recurring time in enrolled patients was compared with the mean time in the literature

CONTACTS AND LOCATIONS:
Overall Officials: Nu Zhang, Professor, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China